CLINICAL TRIAL: NCT03124576
Title: Reappraisal of Atrial Fibrillation: Interaction Between HyperCoagulability, Electrical Remodeling, and Vascular Destabilisation in the Progression of AF- The Tissue Bank Project
Brief Title: Reappraisal of Atrial Fibrillation: RACE-V - Work Package 5
Acronym: RACE V- WP 5
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Ziekenhuis Maastricht (Other)
Responsible Party: Principal Investigator, J. G. Maessen, Prof. Dr., Academisch Ziekenhuis Maastricht
Other Study IDs: NL56796.068.16
Record Dates: First submitted 2016-11-01; First posted 2017-04-24 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — atrial tissue samples, whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- control group: Without history of atrial fibrillation/without newly developed atrial fibrillation detected by continuous rhythm monitoring with a an Implantable loop recorder
  Interventions: Device: Implantable loop recorder
- group B: Patients without history of atrial fibrillation, with new onset atrial fibrillation detected by continuous rhythm monitoring with a an Implantable loop recorder
  Interventions: Device: Implantable loop recorder
- group C: Patients with self-terminating atrial fibrillation at inclusion Implantable loop recorder is used for continuous rhythm monitoring
  Interventions: Device: Implantable loop recorder
- group D: Patients with non-self-terminating atrial fibrillation at inclusion Implantable loop recorder is used for continuous rhythm monitoring
  Interventions: Device: Implantable loop recorder

INTERVENTIONS:
Device: Implantable loop recorder — Continuous rhythm monitoring Medtronic
  Other Names: Reveal LINQ™,Medtronic; ConfirmTM, St. Jude; BiomonitorTM, Biotronik

SUMMARY:
In the proposed study the investigators aim to clarify the relative contribution of these different mechanisms to the progression of atrial fibrillation (AF). Also the contribution of the individual genetic background will be investigated. Furthermore, the investigators aim to identify clinical parameters and biomarkers informing on the main mechanisms of AF progression in atrial tissue.

For this purpose, in all included patients atrial biopsies will be taken during cardiac surgery.

DETAILED DESCRIPTION:
An estimated 380 patients will be included

Four patient categories will be included enabling to study patients with different stages of AF progression;

1. Patients without history of atrial fibrillation, without new onset atrial fibrillation detected by continuous rhythm monitoring after surgery (control group),
2. Patients without history of atrial fibrillation, with new onset atrial fibrillation detected by continuous rhythm monitoring,
3. Patients with self-terminating atrial fibrillation at inclusion, and
4. Patients with non-self-terminating atrial fibrillation at inclusion. At baseline in-depth phenotyping and genotyping will be performed. Continuous rhythm monitoring will also be performed in all patients. The combination of extensive phenotyping, genotyping and atrial fibrillation burden follow-up offers the unique opportunity to study the atrial tissue alterations and atrial gene expression changes in different stages of atrial fibrillation progression and to correlate these data to the phenotype of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Undergoing first elective open chest cardiac surgery or surgical ablation for atrial fibrillation;
* Able and willing to sign informed consent for the registry;
* Able and willing to undergo implantation of implantable loop recorder (unless the patients has a pacemaker or implantable cardioverter-defibrillator (ICD) with atrial leads)

Exclusion Criteria:

* • Deemed unsuitable or not willing to undergo implantation of implantable loop recorder or attend follow-up visits.

  * Pregnancy.
  * Life expectancy of less than 2.5 years.
  * History of prior cardiac surgery or ablation for atrial fibrillation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 380 patiënts undergoing elective open chest heart surgery.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2016-11; Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Biochemical factors in atrial biopsies and blood samples | 2.5 year follow up
  Biochemical factors in atrial biopsies and blood samples associated with atrial fibrillation and contributing to atrial fibrillation progression
Molecular factors in atrial biopsies and blood samples | 2.5 year follow up
  Molecular factors in atrial biopsies and blood samples associated with atrial fibrillation and contributing to atrial fibrillation progression
Genetic factors in atrial biopsies and blood samples | 2.5 year follow up
  Genetic factors in atrial biopsies and blood samples associated with atrial fibrillation and contributing to atrial fibrillation progression

SECONDARY OUTCOMES:
Atrial fibrillation burden | 2.5 year follow up
  Atrial fibrillation burden
Number of atrial fibrillation episodes | 2.5 year follow up
  Number of atrial fibrillation episodes
Duration of atrial fibrillation episodes | 2.5 year follow up
  Duration of atrial fibrillation episodes
Major adverse cardiovascular and cerebrovascular events | 2.5 year follow up
  Major adverse cardiovascular and cerebrovascular events (i.e. death, stroke, myocardial infarction)
First recurrent atrial fibrillation; | 2.5 year follow up
  First recurrent atrial fibrillation
AF progression | 2.5 year follow up
  Self-terminating atrial fibrillation turning into non-self-terminating atrial fibrillation measured from ECGs and implantable loop recorders
AF complexity | 2.5 year follow up
  Electrical atrial fibrillation complexity or signs of atrial conduction disturbances measured from ECGs

CONTACTS AND LOCATIONS:
Overall Officials: Jos Maessen, Prof. Dr., Principal Investigator — Academisch Ziekenhuis Maastricht
Locations (1):
- AZMaastricht, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gilbers MD, Kawczynski MJ, Bidar E, Maesen B, Isaacs A, Winters J, Linz D, Rienstra M, van Gelder I, Maessen JG, Schotten U. Clinical Predictors of Device-Detected Atrial Fibrillation During 2.5 Years After Cardiac Surgery: Prospective RACE V Cohort. JACC Clin Electrophysiol. 2024 May;10(5):941-955. doi: 10.1016/j.jacep.2024.01.013. Epub 2024 Mar 13. PMID 38483418